CLINICAL TRIAL: NCT01671098
Title: Sinonasal Gas Exchange Dynamics The Aerodynamic Theory of the Sinonasal Interface
Brief Title: Sinonasal Gas Exchange Dynamics
Status: Completed | Type: Observational
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Anil Gungor MD, Associate Professor, Louisiana State University Health Sciences Center Shreveport
Other Study IDs: 06301998
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Sinusitis
Keywords: nitric oxide; sinuplasty
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control: Healthy adults
- Balloon Sinuplasty: Patients who had balloon sinuplasty
- FESS-Uncinectomy: Patients who had FESS-Uncinectomy

SUMMARY:
Sinonasal gas exchange is facilitated by the unique anatomy and topography of the sinonasal interface that represents a collection of airfoils creating an aerodynamic structure. The airflow during respiration generates positive and negative pressures that power the gas exchange between the sinuses and the nose. Major surgical alteration of the interface reduces the rate and velocity of the exchange. Minimally invasive procedures aimed at preserving the natural anatomy, topography and aerodynamic configuration of the interface will have negligible effects on sinonasal gas exchange.

ELIGIBILITY:
Inclusion Criteria:

* Control:

  * normal healthy adult volunteers ages 18-65,
* without allergies by history and allergy test,
* non-smoker,
* not using steroids. Study group 1: adult subjects who had maxillary sinus balloon sinuplasty (with intact uncinate and ethmoid complex) Study group 2: adult subjects who had endoscopic maxillary antrostomy and uncinectomy.

Exclusion criteria:

* active acute or chronic infection,
* nasal polyps,
* severe nasal or septal deformity,
* cystic fibrosis,
* systemic illness (diabetes, hypertension etc.),
* vulnerable population (children, pregnant women, institutionalized individuals etc.)
* severe nasal and/or septal deviation,
* hypersensitivity or intolerance to study medications (topical and local anesthetics) any turbinate surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients who had balloon sinuplasty of traditional endoscopic uncinectomy for treatment of chronic maxillary sinusitis
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Sinonasal gas exchange rate | 2 years
  ANALYZE AND DEFINE GAS EXCHANGE PATTERNS IN THE MAXILLARY SINUS DURING NASAL RESPIRATION IN NORMAL SINUSES AND COMPARE WITH SURGICALLY MODIFIED SUBJECTS THAT WILL INCLUDE MAXILLARY SINUSES AFTER ENDOSCOPIC SINUS SURGERY AND BALLOON SINUPLASTY.

SECONDARY OUTCOMES:
NO production rate | 2 years
  ANALYZE AND DEFINE NITRIC OXIDE PRODUCTION RATE AND VARIABLES IN NORMAL AND SURGICALLY ALTERED MAXILLARY SINUSES

CONTACTS AND LOCATIONS:
Overall Officials: Anil A Gungor, MD, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- LSU Health ACC, Shreveport, Louisiana, United States